CLINICAL TRIAL: NCT00269113
Title: A Randomized, Open-label Study of the Effect of MabThera Plus Chemotherapy Versus Chemotherapy Alone on Clinical Response in Patients With Indolent Non-Hodgkin's and Mantle Cell Lymphoma
Brief Title: A Study of MabThera (Rituximab) in Patients With Advanced Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M39023
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Results first posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: rituximab [MabThera/Rituxan]; Drug: Standard chemotherapy
- 2 (Active Comparator)
  Interventions: Drug: Standard chemotherapy

INTERVENTIONS:
Drug: rituximab [MabThera/Rituxan] — 375mg/m2 iv monthly for 8 cycles
  Arms: 1
Drug: Standard chemotherapy — As prescribed

SUMMARY:
This 2 arm study will compare the efficacy and safety of the standard chemotherapy of the East German Study Group for Hematology and Oncology versus standard chemotherapy plus MabThera (375mg/m2 iv, once monthly for 8 cycles) in patients with indolent non-Hodgkin's and mantle cell lymphoma. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* advanced, low-grade non-Hodgkin's and mantle cell lymphoma.

Exclusion Criteria:

* possibility of curative radiation therapy;
* secondary NHL;
* participation in another clinical trial eg with cytostatic chemotherapy or cytokines;
* concomitant diseases and/or restricted organ function precluding therapy according to the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 1998-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (26):
- Germany (26):
  - Berlin
  - Bochum
  - Bonn
  - Borna
  - Chemnitz
  - Cottbus
  - Dresden
  - Dülmen
  - Erfurt
  - Frankfurt (Oder)
  - Greifswald
  - Güstrow
  - Halle
  - Jena
  - Leipzig
  - Magdeburg
  - Marburg
  - Neubrandenburg
  - Nordhausen
  - Potsdam
  - Riesa
  - Rostock
  - Schwerin
  - Stralsund
  - Trier
  - Zella-Mehlis

RESULTS

PARTICIPANT FLOW:
Groups:
- Mitoxantrone, Chlorambucil, Prednisolone (MCP): Participants received mitoxantrone 8 milligrams per square meter (mg/m^2), intravenously (IV), on Days 1 and 2, chlorambucil 3 times (x) 3 mg/m^2, by mouth (PO), every 8 hours on Days 1 through 5, and prednisolone at 25 mg/m^2, PO on Days 1 through 5. This cycle was repeated at 4-week intervals for a minimum of 6 cycles and a maximum of 8 cycles. After Cycles 2 and 6, participants were assessed for response; participants with no change or with progressive disease (or with minimal response at Cycle 6) were withdrawn from therapy. Participants achieving a complete remission (CR) or partial remission (PR) following induction therapy with MCP were administered maintenance therapy (per standard of care and at the discretion of the investigator) with interferon (IFN) alpha 3 x 4.5 million international units (IU) per week, subcutaneously (SC), until progression or withdrawal. Participants could have also received 3 x 500 mg of paracetamol/day during the first weeks of IFN therapy.
- Rituximab + MCP: Participants received rituximab 375 mg/m^2, IV on Day 1, mitoxantrone 8 mg/m^2, IV, on Days 3 and 4, chlorambucil 3 x 3 mg/m^2, PO every 8 hours on Days 3 through 7, and prednisolone 25 mg/m^2, PO on Days 3 through 7. This cycle was repeated at 4-week intervals for a minimum of 6 cycles and a maximum of 8 cycles. After Cycles 2 and 6, participants were assessed for response; participants with no change or with progressive disease (or with minimal response at Cycle 6) were withdrawn from therapy. Participants achieving a CR or PR following induction therapy with MCP were administered maintenance therapy (per standard of care and at the discretion of the investigator) with IFN alpha 3 x 4.5 mIU per week, SC, until progression or withdrawal. Participants could have also received 3 x 500 mg of paracetamol/day during the first weeks of IFN therapy.
Period: Overall Study
Arm/Group | Mitoxantrone, Chlorambucil, Prednisolone (MCP) | Rituximab + MCP
Started | 177 | 183
Completed | 103 | 146
Not Completed | 74 | 37
Not completed — Adverse Event | 14 | 7
Not completed — Lack of Efficacy | 35 | 18
Not completed — Early Improvement | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Death | 6 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Protocol Violation | 15 | 5
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) Population: all participants included in the study, who began a therapy and received at least 1 therapy cycle.
Groups:
- Mitoxantrone, Chlorambucil, Prednisolone (MCP): Participants received mitoxantrone 8 mg/m^2, IV, on Days 1 and 2, chlorambucil 3 x 3 mg/m^2, PO, every 8 hours on Days 1 through 5, and prednisolone at 25 mg/m^2, PO on Days 1 through 5. This cycle was repeated at 4-week intervals for a minimum of 6 cycles and a maximum of 8 cycles. After Cycles 2 and 6, participants were assessed for response; participants with no change or with progressive disease (or with minimal response at Cycle 6) were withdrawn from therapy. Participants achieving a CR or PR following induction therapy with MCP were administered maintenance therapy (per standard of care and at the discretion of the investigator) with IFN alpha 3 x 4.5 mIU per week, SC, until progression or withdrawal. Participants could have also received 3 x 500 mg of paracetamol/day during the first weeks of IFN therapy.
- Total: Total of all reporting groups
Arm/Group | Mitoxantrone, Chlorambucil, Prednisolone (MCP) | Rituximab + MCP | Total
Number analyzed (Participants) | 177 | 181 | 358
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (8.7) | 60.4 (8.3) | 60.4 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 79 | 168
  Male | 88 | 102 | 190

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving CR or PR at the End of Therapy
Description: CR was defined as a complete remission of all objective medical findings at the time of restaging, with complete resolution of pre-existing swelling of the lymph nodes, as well as a pre-existing hepatomegaly and splenomegaly, for at least 4 weeks. This was in exclusion of persistent lymphoma infiltration of the bone marrow by means of bone marrow biopsy; normalization of blood counts with granulocytes greater than (>)1.5 giga particles per liter (Gpt/L) (which is the equivalent of 10^9/L), hemoglobin (Hb) >7.5 millimoles per liter (mmol/L), and platelets less than (<) 100 Gpt/L. PR was defined as greater than or equal to (≥)50 percent (%) reduction of all measurable and evaluable lymphoma manifestations (sum of the products of the 2 largest perpendicular diameters) for at least 4 weeks without occurrence of new manifestations and normalization of blood counts.
Time Frame: Following completion of 6 cycles (24 weeks)
Population: The ITT centroblastic-centrocytic (cbcc)/Follicular Lymphoma (FL) (collectively, ITTcbcc/FL) population included all participants in the ITT population with cbcc lymphoma (target population).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mitoxantrone, Chlorambucil, Prednisolone (MCP) | Rituximab + MCP
Number analyzed (Participants) | 96 | 105
percentage of participants | 75.0 [65.1 to 83.3] | 92.4 [85.5 to 96.7]
Statistical Analysis 1: Comparison: Mitoxantrone, Chlorambucil, Prednisolone (MCP) vs Rituximab + MCP; Test type: Superiority or Other; p = 0.0009, Fisher Exact; Difference in percentage of participants = 17.4, 95% CI 2-sided [6.4 to 28.4]

2. Secondary Outcome: Progression-Free Survival (PFS) - Percentage of Participants Event Free at 24 Months
Description: PFS was defined as the interval from randomization date to progression of disease or death from non-Hodgkin's Lymphoma (NHL). Progression of disease was defined as: increase in the frequency and severity of disease symptoms; occurrence of new nodal or extranodal lymphoma manifestations; volume increase of pre-existing lymphoma manifestations by more than 25%; or increase of splenomegaly by more than 25%. Data were analyzed by means of Kaplan-Meier estimators and log-rank tests at the significance level of alpha equals (=) 5% for difference between the treatment groups.
Time Frame: 24 months
Population: ITTcbcc/FL Population
Measure: Number; unit: percentage of participants
Arm/Group | Mitoxantrone, Chlorambucil, Prednisolone (MCP) | Rituximab + MCP
Number analyzed (Participants) | 96 | 105
percentage of participants | 57.6 | 86.7
Statistical Analysis 1: Comparison: Mitoxantrone, Chlorambucil, Prednisolone (MCP) vs Rituximab + MCP; Test type: Superiority or Other; p < 0.0001, Log Rank

3. Secondary Outcome: Overall Survival (OS) - Percentage of Participants Alive at 24 Months
Description: OS was defined as interval from randomization to date of death of any cause. Data were analyzed by means of Kaplan-Meier estimators and log-rank tests at the significance level of alpha=5% for difference between the treatment groups.
Time Frame: Month 24
Population: ITTcbcc/FL Population
Measure: Number; unit: percentage of participants
Arm/Group | Mitoxantrone, Chlorambucil, Prednisolone (MCP) | Rituximab + MCP
Number analyzed (Participants) | 96 | 105
percentage of participants | 78.8 | 93.7
Statistical Analysis 1: Comparison: Mitoxantrone, Chlorambucil, Prednisolone (MCP) vs Rituximab + MCP; Test type: Superiority or Other; p = 0.0127, Log Rank

4. Secondary Outcome: Event-Free Survival (EFS) - Percentage of Participants Event Free at 24 Months
Description: EFS was defined as the interval from randomization date to therapy failure. Therapy failure was defined after 2 cycles as no change (NC) or progression of disease (PD); after 6 cycles as minimal response [MR], NC, or PD); or death from any cause. NC is defined as tumor regression of <25%, stable disease and progression ≤25%. PD was defined as the increase in the frequency and severity of disease symptoms, occurrence of new nodal or extranodal lymphoma manifestations, volume increase of pre-existing lymphoma manifestations by more than 25%, and increase of splenomegaly by more than 25%. MR was defined as tumor regression between 50% (<50%) and 25% (≥25%) for at least 4 weeks without occurrence of new manifestations. Data were analyzed by means of Kaplan-Meier estimators and log-rank tests at the significance level of alpha=5% for difference between the treatment groups.
Time Frame: Month 24
Population: ITTcbcc/FL Population
Measure: Number; unit: percentage of participants
Arm/Group | Mitoxantrone, Chlorambucil, Prednisolone (MCP) | Rituximab + MCP
Number analyzed (Participants) | 96 | 105
percentage of participants | 50.9 | 83.6
Statistical Analysis 1: Comparison: Mitoxantrone, Chlorambucil, Prednisolone (MCP) vs Rituximab + MCP; Test type: Superiority or Other; p < 0.0001, Log Rank

5. Secondary Outcome: Disease-Free Survival (DFS) - Percentage of Participants Event Free at 24 Months
Description: DFS was defined as the interval from first assessment of CR to PD. PD is an increase in the frequency and severity of disease symptoms, the occurrence of new nodal or extranodal lymphoma manifestations, the volume increase of pre-existing lymphoma manifestations by more than 25%, increase of splenomegaly by more than 25%. Data were analyzed by means of Kaplan-Meier estimators and log-rank tests at the significance level of alpha=5% for difference between the treatment groups.
Time Frame: Month 24
Population: ITTcbcc/FL Population
Measure: Number; unit: percentage of participants
Arm/Group | Mitoxantrone, Chlorambucil, Prednisolone (MCP) | Rituximab + MCP
Number analyzed (Participants) | 96 | 105
percentage of participants | 69.6 | 86.5
Statistical Analysis 1: Comparison: Mitoxantrone, Chlorambucil, Prednisolone (MCP) vs Rituximab + MCP; Test type: Superiority or Other; p = 0.0186, Log Rank

6. Secondary Outcome: Response Duration - Percentage of Participants Event Free at 24 Months
Description: Response duration defined as interval from first assessment of CR/PR to PD. PD is an increase in the frequency and severity of disease symptoms, occurrence of new nodal or extranodal lymphoma manifestations, volume increase of pre-existing lymphoma manifestations by more than 25%, increase of splenomegaly by more than 25%. Data were analyzed by means of Kaplan-Meier estimators and log-rank tests at the significance level of alpha=5% for difference between the treatment groups.
Time Frame: Month 24
Population: ITTcbcc/FL Population
Measure: Number; unit: percentage of participants
Arm/Group | Mitoxantrone, Chlorambucil, Prednisolone (MCP) | Rituximab + MCP
Number analyzed (Participants) | 96 | 105
percentage of participants | 60.3 | 87.7
Statistical Analysis 1: Comparison: Mitoxantrone, Chlorambucil, Prednisolone (MCP) vs Rituximab + MCP; Test type: Superiority or Other; p = 0.0002, Log Rank

7. Secondary Outcome: Time to Next Treatment - Percentage of Participants Who Did Not Need New Treatment at 24 Months
Description: Time to next treatment was defined as the interval from randomization date to the time when new treatment was needed. Data were analyzed by means of Kaplan-Meier estimators and log-rank tests at the significance level of alpha=5% for difference between the treatment groups.
Time Frame: Month 24
Population: ITTcbcc/FL Population
Measure: Number; unit: percentage of participants
Arm/Group | Mitoxantrone, Chlorambucil, Prednisolone (MCP) | Rituximab + MCP
Number analyzed (Participants) | 96 | 105
percentage of participants | 54.6 | 72.0
Statistical Analysis 1: Comparison: Mitoxantrone, Chlorambucil, Prednisolone (MCP) vs Rituximab + MCP; Test type: Superiority or Other; p = 0.0017, Log Rank

ADVERSE EVENTS:
Arm/Group | Mitoxantrone, Chlorambucil, Prednisolone (MCP) | Rituximab + MCP
Serious Adverse Events (participants affected / at risk) | 20/177 | 18/183
Other Adverse Events (participants affected / at risk) | 146/177 | 163/183
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mitoxantrone, Chlorambucil, Prednisolone (MCP) (N=177) | Rituximab + MCP (N=183)
Arterial (Vascular disorders) | 0 | 1
Dysrhythmias (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Ischemia (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 0
Cardiovascular: other (Vascular disorders) | 1 | 0
Venous (Vascular disorders) | 0 | 4
Diarrhea (Gastrointestinal disorders) | 1 | 1
Esophagitis/dysphagia (Gastrointestinal disorders) | 1 | 0
Small bowel (Gastrointestinal disorders) | 0 | 1
Gastrointestinal: other (Gastrointestinal disorders) | 3 | 0
Gastrointestinal (Gastrointestinal disorders) | 1 | 0
Gastritis/Ulcer (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cancer rel. symptoms: other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Second malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Fever (General disorders) | 1 | 0
Lethargy (General disorders) | 1 | 0
Febrile neutropenia (Infections and infestations) | 2 | 6
Allergy (Immune system disorders) | 0 | 1
Hemoglobin (Investigations) | 3 | 2
Blood/marrow: other (Blood and lymphatic system disorders) | 0 | 1
Granulocytes (Investigations) | 1 | 0
Platelets (Investigations) | 3 | 3
White blood count (Investigations) | 6 | 12
Death from within 30 days of treatment (General disorders) | 1 | 1
Mood (Psychiatric disorders) | 0 | 1
Neurologic: other (Nervous system disorders) | 3 | 0
Neurologic pain (Nervous system disorders) | 1 | 0
Osseous: other (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Other (General disorders) | 3 | 0
Infection (Infections and infestations) | 13 | 7
Creatine (Investigations) | 1 | 0
Genitourinary: other (Renal and urinary disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Cerebellar (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mitoxantrone, Chlorambucil, Prednisolone (MCP) (N=177) | Rituximab + MCP (N=183)
Anaemia (Blood and lymphatic system disorders) | 38 | 40
Leukopenia (Blood and lymphatic system disorders) | 108 | 130
Thrombocytopenia (Blood and lymphatic system disorders) | 72 | 76
Constipation (Gastrointestinal disorders) | 10 | 16
Diarrhoea (Gastrointestinal disorders) | 19 | 19
Dyspepsia (Gastrointestinal disorders) | 6 | 19
Nausea (Gastrointestinal disorders) | 35 | 35
Vomiting (Gastrointestinal disorders) | 9 | 13
Chills (General disorders) | 1 | 14
Fatigue (General disorders) | 6 | 13
Pyrexia (General disorders) | 12 | 18
Herpes zoster (Infections and infestations) | 10 | 1
Nasopharyngitis (Infections and infestations) | 16 | 20
Oral herpes (Infections and infestations) | 12 | 9
Urinary tract infection (Infections and infestations) | 13 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 6
Dizziness (Nervous system disorders) | 7 | 12
Headache (Nervous system disorders) | 13 | 14
Initial insomnia (Psychiatric disorders) | 4 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 14
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.